CLINICAL TRIAL: NCT07122089
Title: A Multicenter Open-label, Prospective Study to Evaluate the Efficacy and Safety of SIRT Using Yttrium-90 Glass Microspheres Followed by Durvalumab and Tremelimumab for Treatment of Hepatocellular Carcinoma With Portal Vein Thrombosis
Brief Title: Evaluation of SIRT Followed by Immunotherapy for Treatment of Hepatocellular Carcinoma With Portal Vein Thrombosis
Acronym: IOSPHERE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-3-77-001; 2025-A01081-48 (Other: IDRCB)
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular carcinoma; Immunotherapy; Selective internal radiation therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatocellular carcinoma with portal vein thrombosis and without hepatic spread (Experimental): Patient will receive selective internal radiation therapy and immunotherapy as per standard of care.
  SIRT Administration is direct intra-arterial injection in the hepatic artery to target only liver disease and IO will be performed as describe below:
  * Tremelimumab (Imjudo®): 300 mg IV, one-hour infusion;
  * Durvalumab (Imfinzi®): 1500 mg IV, one-hour infusion every 4 weeks.
  Interventions: Device: Selective Internal Radiotherapy; Drug: Tremelimumab; Drug: Durvalumab

INTERVENTIONS:
Device: Selective Internal Radiotherapy — SIRT will use Yttrium-90 glass-microspheres (TheraSphereTM). SIRT needs two steps: the treatment simulation (diagnostic angiography and scintigraphy of hepatic perfusion with 99mTc-MAA) and the administration (during a therapeutic angiography).
  Other Names: SIRT
Drug: Tremelimumab — Tremelimumab should be done 1 to 3 weeks after SIRT and is administrated according to the Summary of Product Characteristic (SPC).
  Other Names: IMJUDO®
Drug: Durvalumab — After the end of the tremelimumab infusion, patient receive durvalumab then one injection every 4 weeks until further progression upon investigator decision. Also administrated according to the Summary of Product Characteristic (SPC).
  Other Names: Imfinzi®

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common primary liver cancer, being the third leading cause of cancer-related death worldwide, with approximately 745 000 deaths reported annually.

For advanced patients, including patients with tumoral portal vein thrombosis (PVT), most treatment guidelines recommend systemic therapy, either combination immunotherapy (IO) or combination of immunotherapy and anti-angiogenic treatment for first line option.

Results for PVT patients are provided in one trial with a median overall survival of 14.2 months with IO underlying the necessity to improve treatment of PVT patients. Two recent other phase 3 trials also reported positive results for different IO regimen.

Selective internal radiation therapy (SIRT) using yttrium-90 (90Y)-loaded glass microspheres (TheraSphereTM) can be used for patients with early stage to locally advanced HCC including PVT patients without extrahepatic spread (EHS). TheraSphereTM is recognized and is reimbursed in France for PVT patients without EHS, since 2019.Several retrospective studies have shown promising results for PVT patients.

Nowadays use of SIRT in locally advanced HCC is regaining interest based on the results of the randomized DOSISPHERE-01 study including non-operable patients, about 70% with PVT. This randomized Phase II trial using 90Y-loaded microspheres sought was noted the effectiveness of 90Y-loaded microspheres using a personalized dosimetry approach versus a standard dosimetry approach.

The use of a systemic treatment as IO after a locoregional treatment with the strong local debulking effect of SIRT is logical and of interest. Indeed, the most frequent pattern of progression after SIRT is recurrence in an untreated area, including untreated liver or EHS. Patients are then usually referred to IO.

Such kind of therapeutic approach, using SIRT followed by IO has already been evaluated in a phase 2 study using nivolumab after 90Y loaded resin microspheres with promising efficacy without safety deterioration.

The aim of this study is to evaluate SIRT followed by IO used according to their current indications in advanced HCC patient with PVT patients and without EHS.

DETAILED DESCRIPTION:
The study plans to included 80 patients and to treated 72 patients (take into account screen failures and SIRT contraindications).

First, patient will receive SIRT using Yttrium-90 glass microspheres. Immunotherapy with an injection of Tremelimumab followed by Durvalumab must be started 1 to 3 weeks after SIRT.

Durvalumab monotherapy is continued every 4 weeks until disease progression, or toxicity leading to definitive treatment discontinuation, or loss of clinical benefit, or investigator decision, or lost for follow-up or death patient.

Patients are followed prior to the occurrence of progressive disease, within a maximum 18-month period after the initiation IO.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18,
2. ECOG Performance Status 0-1,
3. Histologically proven HCC or noninvasive HCC diagnosis according to LiRADS criteria,
4. HCC with Portal vein involvement (PVT), segmental, sectorial or lobar, evaluated by diagnostic imaging (CT scan or MRI),
5. At least one measurable lesion≥ 10mm using mRECIST criteria evaluated by diagnostic imaging,
6. Tumor involvement <50% of the liver,
7. Hepatic reserve after SIRT ≥ 30% (i.e. hepatic parenchyma not treated with SIRT) evaluated by diagnostic imaging
8. No cirrhosis or Compensated cirrhosis (Child Pugh A, ALBI score 1 or 2),
9. SIRT indication confirmed by a multidisciplinary team meeting (i.e. patient not a candidate for liver resection, thermal ablation, or transplantation at the time of study),
10. Registration with a social security scheme,
11. Written and informed consent of the patient.

Exclusion Criteria:

1. Patient with main PVT (partial or complete),
2. Extrahepatic metastases (patients with EHS), except hilum node < 2 cm,
3. Previous episode of ascites and/or presence of ascites, even if only seen on imaging without clinical detection (except minimum blade only peri-hepatic),
4. Previous episode of hepatic encephalopathy and/or hepatic encephalopathy presence at study entry and/or episodes of encephalopathy (Grade ≥2) within 6 months prior to study inclusion,
5. Pulmonary insufficiency (defined by an arterial oxygen pressure (PaO2) of <60 mmHg, or oxygen saturation (SaO2) of <90% (Roussos & Koutsoukou, 2003) or clinically evident chronic obstructive pulmonary disease (COPD),
6. Medical history of radiation pneumonitis or recent pneumonitis, regardless of causality,
7. Previous HCC therapies:

   1. Any prior systemic treatment for HCC;
   2. More than 2 prior TACE (or embolization), in the area to be treated;
   3. Liver resection or ablation <6 months from end of previous treatment to TheraSphere administration;
   4. Liver ablation <3 months from end of previous treatment to TheraSphere administration.
8. Prior exposure to immune mediated therapy for HCC or other disease, such as other anti-PD-1, anti-PDL-1, anti-PDL-2, anti-CTLA-4, antibodies, etc.
9. Previous liver radiation (external beam radiation therapy (EBRT) or peptide receptor radionuclide therapy (PRRT) or SIRT
10. Inadequate hematological, hepatic and renal functions:

    1. Hemoglobin <8,5 g/dl;
    2. Granulocytes <1500/mm3;
    3. Platelets < 50 000 /mm3;
    4. Bilirubin level ≥35 umol/l;
    5. Albumin <28g/L;
    6. Transaminases > 5 UNL;
    7. Creatinine > 1,5 UNL;
    8. INR>2 (or TP <60%) without anti-coagulation.
11. Any contraindication to angiography or selective visceral catheterization,
12. History of any organ allograft, including bone marrow allo and autograft,
13. History of active primary/acquired immunodeficiency, that makes patients unsuitable for additional immunotherapy in this study (per investigator),
14. Active or prior documented autoimmune or inflammatory disorders (including but not limited to inflammatory bowel disease [e.g. ulcerative colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia;
    2. Patients with hypothyroidism (e.g. following Hashimoto's syndrome) stable on hormone replacement therapy;
    3. Any chronic skin condition that does not require systemic therapy;
    4. Patients with celiac disease controlled by diet alone.
15. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion: Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra-articular injection),
16. In the case of background systemic corticosteroid use, doses of prednisone or its equivalent >10 mg/day,
17. Need for premedication of hypersensitivity reactions with Steroids (e.g. CT scan premedication),
18. History of gastrointestinal bleeding within 42 days prior to study inclusion, active GI bleeding and any bleeding diathesis or coagulopathy that is not correctable by usual therapy or hemostatic agents (e.g. closure device). Patients with known varices that have not bled or which have been clinically addressed can enter the study. No endoscopic exploration is required before study inclusion,
19. Presence of biliary stent or sphincterotomy within one year prior to study inclusion,
20. History of malignancy, other than HCC, within two years, except the condition is one of the following:

    1. Adequately treated carcinoma in situ of the cervix, early squamous cell carcinoma or basal cell carcinoma of the skin, localized prostate cancer, breast ductal carcinoma in situ, or low-grade endometrial carcinoma with no myometrial invasion;
    2. Localized prostate cancer under active surveillance;
    3. Other cancer when there is a negligible risk of recurrence or progression or death (5-year OS rate > 90%).
21. Major surgical procedure (as defined by the Investigator) within 42 days prior to study inclusion,
22. A history of severe allergy or intolerance to contrast agents, narcotics, sedatives, or atropine that cannot be managed medically,
23. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients that cannot be managed medically,
24. Active infection, including:

    1. Tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice),
    2. HBV* and Hep D co-infection,
    3. Human immunodeficiency virus** (HIV 1/2 antibodies) plus HCV or HBV* co-infection.

       * Patients with active HBV infection or HCV infection must be managed according to local standard of care. Patients must show evidence of viral disease stabilization prior to inclusion.

         * Patients with Human Immunodeficiency Virus (HIV) infection are eligible, provided the HIV infection is well controlled with no current or previous AIDS-related complications and CD4+ T-cell (CD4+) counts ≥ 350 cells/µL
25. Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab and/or tremelimumab. Note: patients, if enrolled, should not receive live vaccine whilst receiving durvalumab and/or tremelimumab and up to 30 days after the last dose of durvalumab and/or tremelimumab,
26. Participation in another clinical trial in the 4 weeks prior to enrollment, unless it is an observational study or a 4-week no-treatment follow-up phase of an interventional study,
27. Female patients who are pregnant (a negative serum pregnancy test is mandatory for inclusion) or breastfeeding and who do not want to stop breastfeeding. Male or female patients of reproductive potential who are not willing to employ any effective birth control method from screening and for at least 3 months post the last dose of study treatment (durvalumab ± tremelimumab and/or TheraSphere), whichever is later,
28. Unstable chronic disease or evidence of any disease or condition that would place the patient at undue risk and preclude safe use of TheraSphere, durvalumab and tremelimumab treatment as deemed by the site principal investigator,
29. Patients who are not able to follow the TheraSphere, durvalumab or tremelimumab treatment requirements,
30. Persons deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care under articles L. 3212-1 and L. 3213-1 who are not covered by the provisions of Article L. 1121-8 and persons admitted to a health or social establishment for purposes other than research, including:

    1. Persons receiving psychiatric treatment;
    2. Persons admitted to a health or social establishment for purposes other than research;
    3. Person of full age under curatorship;
    4. Adult subject to a mandate for future protection, a family authorization, or a guardianship measure.

Angiograhy and dosimetry exclusion criteria:

1. Cone Beam CT (CBCT) or Technetium-99m Macro Aggregated Albumin (99mTc-MAA) hepatic arterial perfusion scintigraphy shows any deposition to the gastrointestinal tract that may not be corrected by angiographic techniques,
2. 99mTc-MAA hepatic arterial perfusion scintigraphy shows poor tumor targeting and/or a poor portal vein thrombosis (PVT) targeting (99mTc-MAA uptake ≤ normal liver uptake),
3. The dosimetry endpoints cannot be reached (refer to the supplement A "TheraSphere Treatment Planning, Dosimetry Guidance document"),
4. Shunting of blood to the lungs that could result in delivery of >30 Gy to the lungs in a single treatment, or >50 Gy cumulative dose to the lungs in case of multiple TheraSphere treatments, as seen on 99mTc-MAA hepatic arterial perfusion scintigraphy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2030-01-02 (Estimated); Study Completion 2030-01-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, an average of 4 years
  The Objective Response Rate (ORR) is defined as the proportion of patients who have either a Partial Response (PR) or a Complete Response (CR) to treatment. CR and PR are the best overall response across all time points of tumor evaluation. Overall tumor response at each time point is assessed according to the modified RECIST criteria for HCC.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Garin, MD PHD, Principal Investigator — Centre de Lutte Contre Le cancer Eugène Marquis